CLINICAL TRIAL: NCT04490005
Title: Outcome pRognostication of Acute Brain Injury With the NeuroloGical Pupil
Brief Title: Outcome pRognostication of Acute Brain Injury With the NeuroloGical Pupil indEx
Acronym: ORANGE
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: University of Lausanne (Other); Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Other Study IDs: ORANGE
Record Dates: First submitted 2020-07-01; First posted 2020-07-28 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Acute Brain Injury; Pupillary Reflex Impaired
Keywords: acute brain injury; pupillometry; intracranial hypertension; neurological outcome
MeSH Terms: conditions — Brain Injuries; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Acute brain injury: Intensive care unit (ICU) admission after ABI, including traumatic brain injury (TBI), aneurysmal subarachnoid haemorrhage (SAH) and intracerebral haemorrhage (ICH)
  • Age 18 years old.
  Interventions: Other: pupillometry

INTERVENTIONS:
Other: pupillometry — evaluation of pupillary reflex by using the Neuroptics Pupillometer every 4 hours during ICU stay

SUMMARY:
The use of quantitative, automated, infrared technology for pupillary examination has long been used in ophthalmology and anesthesiology research. Its interest in neurocritical care has progressively grown, in parallel with the advancements in device technology. In this regard, the use of the noninvasive NPi®-200 pupillometer (Neuroptics, Laguna Hills, California, USA) allows the measurement of a series of dynamic pupillary variables (including the percentage pupillary constriction, latency, constriction velocity, and dilation velocity), which can be integrated into an algorithm, to compute the Neurological Pupil index (NPi). The NPi is a proprietary scalar index with values between 0 and 5 (with a 0.1 decimal precision), an NPi value < 3 indicating an abnormal pupillary reactivity. Importantly, the NPi is not influenced by sedation-analgesia, at the doses used in neurocritical care practice, and by mild hypothermia.

Preliminary single-center data recently demonstrated that abnormal NPi is associated with worse outcome in patients with traumatic and hemorrhagic ABI, and can be a useful adjunct for ICP monitoring and therapy. There is currently a great need for quantitative tools to predict early prognostication in ABI patients, and the NPi appears of potential great value.

We hypothesize that:

1. Abnormal NPi (defined as NPi <3) are strongly predictive of poor GOS-E (1-4) at 6 months after the acute event.
2. NPi=0 is strongly predictive of mortality (GOS 1).
3. Abnormal NPi is predictive of a higher ICP 20 index (number of end-hourly measures of ICP >20 mm Hg divided by the total number of measurements, multiplied by 100) and a greater burden of interventions needed to control ICP (measured by the Therapy Intensity Level scale for ICP management, Therapy Intensity Level (TIL) 4).

Methods This international multicentre prospective observational study aims to recruit >400 patients admitted to intensive care units.

Duration of the study 18 months, including 12-month of recruitment based on 60 patients/centre plus 6 months GOS-E follow-up.

DETAILED DESCRIPTION:
Introduction Pupillary examination, and in particular pupillary light reactivity (PLR), is fundamental for intensive care unit (ICU) monitoring and follow-up of patients with acute brain injury (ABI), and has both diagnostic and prognostic values. Secondary cerebral insults, e.g. elevated intracranial pressure (ICP) may alter midbrain function and cause abnormalities in pupil size, symmetry and PLR. Sustained or newfound pupillary abnormalities are associated with a worse outcome, and indeed PLR is a robust validated predictor in several prognostic models, such as the CRASH (Corticosteroid Randomization after Significant Head Injury) and the IMPACT (International Mission for Prognosis and Analysis of Clinical Trials) scores. In current clinical practice however, pupillary examination is performed using a manual, hand-held light source (e.g. pen torch), implying that the evaluation of pupillary size and reactivity remains essentially based on a visual qualitative assessment. This traditional approach has several limitations, such as limited precision (especially in patients with small pupil size), significant intra- and inter-observer variability, differences in ambient light exposure between measurements, or the technique used to direct the stimulus (i.e. intensity, proximity, duration and orientation of the light source).

The use of quantitative, automated, infrared technology for pupillary examination has long been used in ophthalmology and anesthesiology research. Its interest in neurocritical care has progressively grown, in parallel with the advancements in device technology. In this regard, the use of the noninvasive NPi®-200 pupillometer (Neuroptics, Laguna Hills, CA, USA) allows the measurement of a series of dynamic pupillary variables (including the percentage pupillary constriction, latency, constriction velocity, and dilation velocity), which can be integrated into an algorithm, to compute the Neurological Pupil index (NPi). The NPi is a proprietary scalar index with values between 0 and 5 (with a 0.1 decimal precision), an NPi value < 3 indicating an abnormal pupillary reactivity. Importantly, the NPi is not influenced by sedation-analgesia, at the doses used in neurocritical care practice, and by mild hypothermia.

Preliminary single-center data recently demonstrated that abnormal NPi is associated with worse outcome in patients with traumatic and hemorrhagic ABI, and can be a useful adjunct for ICP monitoring and therapy. There is currently a great need for quantitative tools to predict early prognostication in ABI patients, and the NPi appears of potential great value. For this purpose, large multicenter studies are required. The Investigators recently conducted an international multicenter study that demonstrated the prognostic value of NPi in the setting of early prognostication of ABI following cardiac arrest. Here, the Investigators aim at evaluating the prognostic value of the NPi in patients with ABI following traumatic brain injury (TBI), aneurysmal subarachnoid hemorrhage (SAH) or intracerebral hemorrhage (ICH) at risk of secondary ICP elevation.

Research questions

The Investigators hypothesize that:

1. Abnormal NPi (defined as NPi <3) are strongly predictive of poor GOS-E (1-4) at 6 months after the acute event.
2. NPi=0 is strongly predictive of mortality (GOS 1).
3. Abnormal NPi is predictive of a higher ICP 20 index (number of end-hourly measures of ICP >20 mm Hg divided by the total number of measurements, multiplied by 100) and a greater burden of interventions needed to control ICP (measured by the Therapy Intensity Level scale for ICP management, TIL 4).

Methods

Prospective, observational, international cohort study focused at identifying the relationship of NPi with:

* long-term outcome defined as 6-months mortality and neurological recovery, measured with the extended Glasgow Outcome Score, GOS-E;
* intracranial hypertension.

Sample size calculation No formal sample size calculation has been performed due to the exploratory nature of the study. However, the Investigators expect to recruit a total of 420 patients, 140 per pathology for whom GOSE will be performed (i.e. TBI, ICH, SAH), over a 12-months period. Therefore, the twelve participating centres will contribute, based on their potentiality of recruitment, with a minimum of 20 patients.

Screening All patients admitted to the participating ICUs in coma after ABI will be screened daily and entered into a screening log . Each ICU will recruit eligible patients for 12 consecutive months and collect data for each recruited patient daily in an expanded electronic case report form (eCRF). Both common-data elements and etiology-specific data will be collected.

Demographics and Medical History Demographic characteristics and medical history information will be extracted from patients' medical records including gender, age, co-morbidities, diagnosis, timeline and clinical presentation of acute brain injury. All NPi and ICP monitoring data, as well as additional neuro-monitoring and neuroimaging data will be extracted from patients' medical records too and documented in the eCRF.

NPi Data and Daily eCRF The daily eCRF Data Capture will be completed for NPi (collected every 4 hours) and for ICP (matched to NPi), every day, from admission up to day 7 . Data collected will also include additional ICP derived variables and interventions.

Outcome measures Glasgow Outcome Scale-Extended (GOS-E) as main outcome will be collected at ICU/hospital discharge and at 6 months). Data on the cause of death will be collected as well. The GOS-E at the End-of-Study will be collected via telephone-structured interviews to patients and/or family members using a validated questionnaire.

Statistical methods No formal sample size calculation has been performed due to the exploratory nature of the study. However, the Investigators expect to recruit a total of 420 patients, 140 per pathology (i.e. TBI, ICH, SAH), over a 12-months period.

Therefore, the twelve participating centres will contribute, based on their potentiality of recruitment, with a minimum of 20 patients.

Data will be summarised by counts and percentages and quartiles or means and standard deviation, as appropriate, for qualitative and quantitative characteristics, respectively.

Unsupervised and supervised methods will be applied with explorative purposes using the individual NPi longitudinal measurements. For example, the pattern recognition of longitudinal profiles and the cluster trajectory analyses will be used in order to identify patterns of NPi trajectories associated with prognosis. NPi trends will be also described graphically and modelled by longitudinal mixed models using splines.

A Cox and a logistic model will be then applied to evaluate the association between the NPi process with the 6-month mortality and the neurological recovery (GOSE≤4 vs GOSE>4) at 6 months, respectively. This will be done considering NPi in categories identifying different potential patterns in NPi profiles or using summary measures that have been already introduced in this context, such as the percentage of NPi<3 observed in the time interval of observation or the area under the trajectory in time. The two eyes will contribute to these analyses with the worst result. This analysis will be done overall on a multivariable model that will also explore a potential interaction effect with the different pathologies, while the improvement with respect to the standard risk factors (e.g. the components of the IMPACT model for TBI patients) will be evaluated by multivariable models on each of the three specific pathologies.

Lastly, the association between NPi and mortality will be evaluated by the use of shared frailty joint models, in which NPi trend in left and right eye will be evaluated by a multivariate mixed model, which outcome will be used to model mortality. Model-based mortality prediction will be computed based on individual NPi trends. The same kind of approach will be used for the binary outcome.

Potential Risks and Benefits Risks The ORANGE study is observational. It does not introduce any interventional procedure. The data is extracted from the patients' medical records and does not affect local standard of care. Hence, the study does not add any interventional risk to the patients recruited.

Confidentiality breach is a potential risk, which will be addressed by patients' data codification. A unique code will be generated by the e-CRF and allocated to every site and every enrolled patient.

Benefits No individual benefit is expected for the study participants. Nevertheless, the results of the study could possibly help us improving the knowledge for a better medical care for similar patients in the future and the generation of hypotheses for further collaborative research.

Data Collection ICUs willing to participate will register electronically and collect data via an electronic Case-Report Form (RedCAP platform). An online training module will be developed to help data collectors in completing the study eCRF. Data collection will be web based, permitting conditional Data Collection screens, i.e. data collectors will be automatically guided as to which sections to complete based on data entered indicating whether Inclusion Criteria are met.

Ethical standards This study is conducted in compliance with the protocol version 3.0 , the current version of the Declaration of Helsinki, the ICH-Good Clinical Practice (GCP) guidelines, as well as local relevant legal and regulatory requirements of every site.

Ethics committee Each investigator will notify the relevant ethics committee, in compliance with the local legislation and rules.

The approval of the protocol (if required by local authorities) must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the 3 chief investigators before the changes are implemented to the study.

Lack of capacity and Delayed Consent Patients recruited in this study will not be able to provide informed consent at the time of recruitment. The responsible clinical/research staff will act as Consultee and consent eligible patients after discussion with the next-of-kin.

If the patient has a Power of Attorney or a Legal tutor or an, he/she will act as Consultee and will be asked to consent/decline participation to the study on legal behalf of the patient.

If patients have Advance Decision Plan including participation in research studies the Plan will be respected and recruitment pursued/abandoned accordingly.

At follow-up, patients who have regained capacity will be asked to provide Informed Consent and will be given the possibility to:

* Provide Informed Consent for the acute data and follow-up.
* Deny research participation and request destruction of acute data collected.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit (ICU) admission after ABI, including traumatic brain injury (TBI), aneurysmal subarachnoid haemorrhage (SAH) and intracerebral haemorrhage (ICH)
* Age > 18 years old.
* Pupillometry available as standard evaluation tool.

Exclusion Criteria:

* ABI not admitted to the ICU.
* Facial trauma not allowing pupils' evaluation.
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No formal sample size calculation has been performed due to the exploratory nature of the study. However, we expect to recruit a total of 420 patients, 140 per pathology for whom GOSE will be performed (i.e. TBI, ICH, SAH), over a 12-months period. Therefore, the six participating centres will contribute, based on their potentiality of recruitment, with a minimum of 20 patients for each of the three pathologies, for a total of 60.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Correlation between abnormal Neurological Pupil index (NPi) and long-term outcome | 6 months
  To evaluate the association between abnormal Neurological Pupil index (NPi) and long-term outcome (6-month mortality and neurological recovery, measured with the extended Glasgow Outcome Score, GOS-E) in patients with ABI.

SECONDARY OUTCOMES:
Correlation between intracranial hypertension and abnormal NPI values | 6 months
  The secondary aim, in patients with ICP monitoring, is to evaluate the relationship of abnormal NPi and intracranial hypertension in order to prognosticate a poor neurological outcome (Glasgow Outcome Scale-Extended)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, MD, Prof, Principal Investigator — University of Milano Bicocca
Locations (14):
- United States (4):
  - Department of Neurology, University of California, San Francisco, California
  - Parnassus Hospital UCSF, San Francisco, California
  - John Hopkins, Baltimore, Maryland
  - Harborview Medical Center, Seattle, Washington
- Erasme Hospital, Université Libre de Bruxelles, Brussels, Belgium
- Department Anesthesia and Critical Care, University Hospital, Grenoble, France
- Universitätsklinikum, Erlangen, Germany
- Italy (3):
  - Spedali Civili, Brescia, BS
  - ASST-MONZA San Gerardo Hospital, Monza, MB
  - Policlinico Gemelli, Roma, RM
- Oslo Universitary Hospital, Oslo, Norway
- Spain (2):
  - Ramón Y Cajal University Hospital, Madrid
  - Hospital Clinic Universitari de València, University of Valencia, Valencia
- Centre Hospitalier Universitaire Vaudois (CHUV), University Hospital and University of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No
Access to data The University of Milano-Bicocca has the property of all the data collected. The data resides at the University Milano-Bicocca as study Sponsor; all procedures will comply with the European Union (EU) regulation on data protection 2016/679 on the protection of natural persons regarding personal data processing and movement. Local site data will be co-owned by each participating centre, and they will be given access to local data for any scientific purpose upon request. By entering data into the ORANGE study database, each centre agrees that the chief can use these data for scientific purposes. Any requests for the use of the data set for subsequent studies will be made to the ORANGE study chief investigators. Any requests for the use of the data set for subsequent studies will be made to the ORANGE study chief investigators.

REFERENCES:
- [Result] Sharshar T, Citerio G, Andrews PJ, Chieregato A, Latronico N, Menon DK, Puybasset L, Sandroni C, Stevens RD. Neurological examination of critically ill patients: a pragmatic approach. Report of an ESICM expert panel. Intensive Care Med. 2014 Apr;40(4):484-95. doi: 10.1007/s00134-014-3214-y. Epub 2014 Feb 13. PMID 24522878
- [Result] Chen JW, Gombart ZJ, Rogers S, Gardiner SK, Cecil S, Bullock RM. Pupillary reactivity as an early indicator of increased intracranial pressure: The introduction of the Neurological Pupil index. Surg Neurol Int. 2011;2:82. doi: 10.4103/2152-7806.82248. Epub 2011 Jun 21. PMID 21748035
- [Result] Chen JW, Vakil-Gilani K, Williamson KL, Cecil S. Infrared pupillometry, the Neurological Pupil index and unilateral pupillary dilation after traumatic brain injury: implications for treatment paradigms. Springerplus. 2014 Sep 23;3:548. doi: 10.1186/2193-1801-3-548. eCollection 2014. PMID 25332854
- [Result] Larson MD, Behrends M. Portable infrared pupillometry: a review. Anesth Analg. 2015 Jun;120(6):1242-53. doi: 10.1213/ANE.0000000000000314. PMID 25988634
- [Result] Larson MD, Singh V. Portable infrared pupillometry in critical care. Crit Care. 2016 Jun 22;20(1):161. doi: 10.1186/s13054-016-1349-7. PMID 27329287
- [Result] Volpi PC, Robba C, Rota M, Vargiolu A, Citerio G. Trajectories of early secondary insults correlate to outcomes of traumatic brain injury: results from a large, single centre, observational study. BMC Emerg Med. 2018 Dec 5;18(1):52. doi: 10.1186/s12873-018-0197-y. PMID 30518336
- [Result] Han J, King NK, Neilson SJ, Gandhi MP, Ng I. External validation of the CRASH and IMPACT prognostic models in severe traumatic brain injury. J Neurotrauma. 2014 Jul 1;31(13):1146-52. doi: 10.1089/neu.2013.3003. Epub 2014 May 12. PMID 24568201
- [Result] Couret D, Boumaza D, Grisotto C, Triglia T, Pellegrini L, Ocquidant P, Bruder NJ, Velly LJ. Reliability of standard pupillometry practice in neurocritical care: an observational, double-blinded study. Crit Care. 2016 Mar 13;20:99. doi: 10.1186/s13054-016-1239-z. PMID 27072310
- [Result] Couret D, Simeone P, Freppel S, Velly L. The effect of ambient-light conditions on quantitative pupillometry: a history of rubber cup. Neurocrit Care. 2019 Apr;30(2):492-493. doi: 10.1007/s12028-018-0664-z. No abstract available. PMID 30604030
- [Result] Olson DM, Stutzman S, Saju C, Wilson M, Zhao W, Aiyagari V. Interrater Reliability of Pupillary Assessments. Neurocrit Care. 2016 Apr;24(2):251-7. doi: 10.1007/s12028-015-0182-1. PMID 26381281
- [Result] Hall CA, Chilcott RP. Eyeing up the Future of the Pupillary Light Reflex in Neurodiagnostics. Diagnostics (Basel). 2018 Mar 13;8(1):19. doi: 10.3390/diagnostics8010019. PMID 29534018
- [Result] Larson MD, Sessler DI. Pupillometry to guide postoperative analgesia. Anesthesiology. 2012 May;116(5):980-2. doi: 10.1097/ALN.0b013e318251d21b. No abstract available. PMID 22433239
- [Result] Morelli P, Oddo M, Ben-Hamouda N. Role of automated pupillometry in critically ill patients. Minerva Anestesiol. 2019 Sep;85(9):995-1002. doi: 10.23736/S0375-9393.19.13437-2. Epub 2019 Mar 29. PMID 30938123
- [Result] Shoyombo I, Aiyagari V, Stutzman SE, Atem F, Hill M, Figueroa SA, Miller C, Howard A, Olson DM. Understanding the Relationship Between the Neurologic Pupil Index and Constriction Velocity Values. Sci Rep. 2018 May 3;8(1):6992. doi: 10.1038/s41598-018-25477-7. PMID 29725074
- [Result] Jahns FP, Miroz JP, Messerer M, Daniel RT, Taccone FS, Eckert P, Oddo M. Quantitative pupillometry for the monitoring of intracranial hypertension in patients with severe traumatic brain injury. Crit Care. 2019 May 2;23(1):155. doi: 10.1186/s13054-019-2436-3. PMID 31046817
- [Result] Aoun SG, Stutzman SE, Vo PN, El Ahmadieh TY, Osman M, Neeley O, Plitt A, Caruso JP, Aiyagari V, Atem F, Welch BG, White JA, Batjer HH, Olson DM. Detection of delayed cerebral ischemia using objective pupillometry in patients with aneurysmal subarachnoid hemorrhage. J Neurosurg. 2020 Jan 1;132(1):27-32. doi: 10.3171/2018.9.JNS181928. Epub 2019 Jan 11. PMID 30641848
- [Result] Osman M, Stutzman SE, Atem F, Olson D, Hicks AD, Ortega-Perez S, Aoun SG, Salem A, Aiyagari V. Correlation of Objective Pupillometry to Midline Shift in Acute Stroke Patients. J Stroke Cerebrovasc Dis. 2019 Jul;28(7):1902-1910. doi: 10.1016/j.jstrokecerebrovasdis.2019.03.055. Epub 2019 Apr 25. PMID 31031146
- [Result] Ong C, Hutch M, Barra M, Kim A, Zafar S, Smirnakis S. Effects of Osmotic Therapy on Pupil Reactivity: Quantification Using Pupillometry in Critically Ill Neurologic Patients. Neurocrit Care. 2019 Apr;30(2):307-315. doi: 10.1007/s12028-018-0620-y. PMID 30298336
- [Result] Phillips SS, Mueller CM, Nogueira RG, Khalifa YM. A Systematic Review Assessing the Current State of Automated Pupillometry in the NeuroICU. Neurocrit Care. 2019 Aug;31(1):142-161. doi: 10.1007/s12028-018-0645-2. PMID 30484008
- [Result] Oddo M, Sandroni C, Citerio G, Miroz JP, Horn J, Rundgren M, Cariou A, Payen JF, Storm C, Stammet P, Taccone FS. Quantitative versus standard pupillary light reflex for early prognostication in comatose cardiac arrest patients: an international prospective multicenter double-blinded study. Intensive Care Med. 2018 Dec;44(12):2102-2111. doi: 10.1007/s00134-018-5448-6. Epub 2018 Nov 26. PMID 30478620
- [Result] Zuercher P, Groen JL, Aries MJ, Steyerberg EW, Maas AI, Ercole A, Menon DK. Reliability and Validity of the Therapy Intensity Level Scale: Analysis of Clinimetric Properties of a Novel Approach to Assess Management of Intracranial Pressure in Traumatic Brain Injury. J Neurotrauma. 2016 Oct 1;33(19):1768-1774. doi: 10.1089/neu.2015.4266. Epub 2016 Feb 11. PMID 26866876
- [Result] Wilson L, von Steinbuechel N, Menon DK, Maas AIR. Outcome assessment after traumatic brain injury - Authors' reply. Lancet Neurol. 2018 Apr;17(4):299-300. doi: 10.1016/S1474-4422(18)30045-0. Epub 2018 Mar 13. No abstract available. PMID 29553376
- [Derived] Petrosino M, Gouvea Bogossian E, Rebora P, Galimberti S, Chesnut R, Bouzat P, Oddo M, Taccone FS, Citerio G; ORANGE Participants and Investigators. Neurological Pupil Index and Intracranial Hypertension in Patients With Acute Brain Injury: A Secondary Analysis of the ORANGE Study. JAMA Neurol. 2025 Feb 1;82(2):176-184. doi: 10.1001/jamaneurol.2024.4189. PMID 39652324
- [Derived] Oddo M, Taccone FS, Petrosino M, Badenes R, Blandino-Ortiz A, Bouzat P, Caricato A, Chesnut RM, Feyling AC, Ben-Hamouda N, Hemphill JC, Koehn J, Rasulo F, Suarez JI, Elli F, Vargiolu A, Rebora P, Galimberti S, Citerio G; ORANGE study investigators. The Neurological Pupil index for outcome prognostication in people with acute brain injury (ORANGE): a prospective, observational, multicentre cohort study. Lancet Neurol. 2023 Oct;22(10):925-933. doi: 10.1016/S1474-4422(23)00271-5. Epub 2023 Aug 28. PMID 37652068
- [Derived] Oddo M, Taccone F, Galimberti S, Rebora P, Citerio G; Orange Study Group. Outcome Prognostication of Acute Brain Injury using the Neurological Pupil Index (ORANGE) study: protocol for a prospective, observational, multicentre, international cohort study. BMJ Open. 2021 May 11;11(5):e046948. doi: 10.1136/bmjopen-2020-046948. PMID 33980528